CLINICAL TRIAL: NCT02724722
Title: Family-based Childhood Behavior Intervention to Decrease Environmental Melamine and Phthalate Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Tsang Wu, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMU-TP103A23
Record Dates: First submitted 2015-03-10; First posted 2016-03-31 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Children and Their Main-care Giver
Keywords: melamine; phthalate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): a simple flyer in one empty bag with face-to-face health education
  Interventions: Behavioral: Assigned intervention
- No Intervention (Placebo Comparator): a simple flyer in one empty bag with no face-to-face health education
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Assigned intervention — a simple flyer plus face-to-face health education and give one bag containing stainless steel-made tableware for eating out use
  Arms: Intervention
Behavioral: No intervention — a simple flyer only with no face-to-face health education and give one bag not containing stainless steel-made tableware for eating out use
  Arms: No Intervention

SUMMARY:
Melamine and phthalates are environmental emerging chemicals, which are ubiquitously present in the public and easily contacted by children through air, foods, and skin. This study aims to examine whether the use of family-based behavior intervention by providing simple flyers plus face-to-face health education point-by-point and give one bag containing stainless steel-made tableware for eating out use to study children's mothers or main-care givers can significantly decrease melamine and phthalates exposure by measuring urinary melamine and metabolites of phthalates (especially DEHP metabolites) in study children and their mothers or main-care givers, when compared to those provided simple flyers only.

DETAILED DESCRIPTION:
Study subjects: Between May 31 and June 17, 2011, 108 children visited the special Phthalates Clinic for Children (PCC) at Kaohsiung Medical University Hospital (KMUH). Thirteen children whose age was older than 10 years, one girl with a history of hormone (leuprorelin) treatment, and thirty-four whose parents did not sign informed consents were excluded. The rest of 60 children are eligible to participate in this study. Because 37 out of the 60 potential study children did provide enough urine for the analyses of phthalates metabolites in our previous study [Wu et al., 2013a; Wu et al., 2013b], in this study, the investigators focus on the 37 study children. After the contact by phone, 24 study children and their mothers or main-care givers are willing to participate in this study intervention.

Study protocol: This is a family-based randomized intervention. The investigators will conduct this study for 2 weeks follow up. The investigators randomly assign 12 study children and their main-care givers (i.e., mothers or grandmothers) to a intervention group and another 12 to a control group. Intervention group means study children and their main-care givers (i.e., mothers or grandmothers) will receive face-to-face health education, besides provided the simple flyers and give one bag containing stainless steel-made tableware for eating out use, how to avoid environmental exposure to melamine and phthalate chemicals based on the evidence-based data from the investigators' laboratory and other researchers. The investigators only provide the simple flyers in a empty bag to the control group. The investigators will collect two one-spot urine samples from two consecutive mornings of the study children and their main-care givers, usually mother or grandmothers, at the baseline. Blood samples of the children were also collected measurement of endocrine profile, including TSH, T4, FT4, T3, and E2. After 2 weeks, another two one-spot urine samples from two consecutive mornings of the study investigators will collect two one-spot urine samples from two consecutive mornings of the study children and their main-care givers, usually mother or grandmothers, every 3 months for analyses.

ELIGIBILITY:
Inclusion Criteria:

* 3-18-yrs healthy children and their main-care givers (i.e., mothers or grandmothers)

Exclusion Criteria:

* Children with any hormone treatment or major chronic diseases such as cancer

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
urinary excretion of melamine | 2 weeks
urinary excretion of five DEHP metabolites (MEHP, 5OH-MEHP, 5oxo-MEHP, 5carboxy-MEPP, and 2carboxy-MMHP) | 2 weeks

SECONDARY OUTCOMES:
oxidative stress markers (8-OHdG, MDA) | 6 months
other six phthalate metabolites of MnBP, MiBP, MEP, MBzP, MMP, and MiNP | 2 weeks
oxidative stress markers (8-OHdG, MDA) | one year
renal injury markers (NAG, microalbumin, beta-2-microglobulin) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsang Wu, MD, ScD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Background] Wu MT, Wu CF, Chen BH, Chen EK, Chen YL, Shiea J, Lee WT, Chao MC, Wu JR. Intake of phthalate-tainted foods alters thyroid functions in Taiwanese children. PLoS One. 2013;8(1):e55005. doi: 10.1371/journal.pone.0055005. Epub 2013 Jan 30. PMID 23383031
- [Background] Wu CF, Chen BH, Shiea J, Chen EK, Liu CK, Chao MC, Ho CK, Wu JR, Wu MT. Temporal changes of urinary oxidative metabolites of di(2-ethylhexyl)phthalate after the 2011 phthalate incident in Taiwanese children: findings of a six month follow-up. Environ Sci Technol. 2013 Dec 3;47(23):13754-62. doi: 10.1021/es403141u. Epub 2013 Nov 18. PMID 24191740